CLINICAL TRIAL: NCT05043961
Title: Determination of the Success Rate of the Palisade Lateral Branch Technique Using Multi-tined Needles for Sacro-iliac Joint Radiofrequency Ablation
Brief Title: Palisade Lateral Branch Technique Using Multi-tined Needles for Sacro-iliac Joint Radiofrequency Ablation
Acronym: TriPal
Status: Terminated | Type: Observational
Why Stopped: Not enough study participants
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Principal Investigator, Maisonneuve-Rosemont Hospital
Other Study IDs: 2022-2704
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sacroiliac; Backache; Chronic Pain
Keywords: radiofrequency ablation; Sacroiliac joint pain; chronic pain
MeSH Terms: conditions — Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Patients who report >50% pain relief after an intra articular sacroiliac joint injection but lasting less than 3 months who are scheduled to receive a SIJ RFA at the Maisonneuve-Rosemont Hospital's Chronic Pain Clinic and who meet inclusion criteria will be offered to participate in this study.
  Intervention:
  Sacroiliac joint rafiofrequency ablation using the bipolar palissade approach and 3-tined needles
  Interventions: Procedure: Palisade sacroiliac joint radiofrequency ablation using 3-tined needles

INTERVENTIONS:
Procedure: Palisade sacroiliac joint radiofrequency ablation using 3-tined needles — Palisade-RF is performed using a conventional temperature-controlled RF generator generating monopolar and bipolar lesions at 85°C for 150 sec, with a 60 sec ramp time. Four, 18 Gauge 3-tined, 90 mm cannulas with an active tip of 10 mm (RF Trident; Diros Technology) will be used along with a four-output radiofrequency generator configured for quadripolar and bipolar output.
  The RF energy is delivered, making one quadripolar or two bipolar lesions at a time. This procedure is repeated at the remaining target sites by leapfroging the needles, until the entire length is lesioned.
  Lesioning the L5 dorsal ramus:
  o The RF needle is inserted at the inflexion between the ala of the sacrum and the S1 superior articular process. The RF energy is delivered, creating a monopolar lesion.

SUMMARY:
The sacro-iliac joint is a large joint that can be the source of chronic pain. Many treatment options have been proposed to treat SIJ pain, with variable efficacy. The next step in managing those patients who can't get sustained pain relief from conservative treatment is radiofrequency ablation (RFA) of the SIJ's posterior innervation.

However, the success rate of SIJ RFA, as determined by the proportion of patients reporting greater than 50% pain relief 6 months after the intervention, varies substantially across studies, ranging from 38-71 %. This may be explained partly by the fact that there may be incomplete lesioning of the target nerves supplying the joint. To overcome these particularities, two RFA techniques have emerged: cooled RFA and bipolar RFA.

Cooled radiofrequency is the one that has been studied the most, and good evidence supports its efficacy. However, its superiority to conventional RF for the treatment of SIJ pain is not confirmed.

Alternatively, a bipolar RFA technique using conventional radiofrequency needles and equipment can be used. The efficacy of this relatively newer technique has been demonstrated by only one study, and although the results were promising, it is not known whether they could be replicated. The success of the palisade technique could be enhanced by using multi-tined expandable electrodes, such as the 3-tined Trident cannulas, with only small increases in cost.

In clinical practice, the palisade technique using 3-tines needles is routinely used. However, its efficacy has not been formally evaluated. The primary objective of this prospective cohort study will be to determine the success rate of the palisade SIJ RFA (P-RF) technique using the 3-tined needles, determined as the proportion of patients reporting >50% pain relief, 6 months after the procedure.

DETAILED DESCRIPTION:
Single center, prospective cohort study. all patients presenting to the Maisonneuve-Rosemont's Pain center with chronic low back pain of SIJ origin who are candidates for SIJ RFA during a two year period will be invited to participate in this study. SIJ RFA will be performed using the palisade technique using 3-tined needles. The patients will be followed for a period of 10 months to determine pain relief, opioid use, satisfaction and impact on disability.

Study design: Prospective, cohort study Population: Patients who are scheduled to receive a SIJ RFA at the Maisonneuve-Rosemont Hospital's Chronic Pain Clinic Duration of study: 2 years Patient included in the study will be followed up for 10 months. Sample size: Approximately 30 patients (anticipated)

General Study procedure This study's methodology will follow the standard practice for treating patients with SIJ pain at the Maisonneuve-rosemont Hospital First, an intraarticular SIJ injection of local anesthetic with a corticosteroid is offered to patients presenting with pain of presumed SIJ origin (predominantly axial low back pain, below the L5 vertebrae, positive SIJ provocation maneuvers). Patients who experience significant pain relief but lasting less than 3 months are offered a SLBB. According to standard practice, all patients receiving a SLBB file a pain diary that evaluates the pain intensity over a 36h period following the block (see Annex 1). This diary is sent back by e-mail to the treating physician and will be deemed positive if >50% pain relief is reported for at least 2h but lasting less than 24h. Patients with a positive SLBB are always considered for SIJ RFA. Patients with a negative SLBB may or may not undergo SIJ RFA, depending on the treating physician. Indeed, although SLBB have been suggested as a more appropriate method for selecting patients who should undergo SIJ RFA, its predictive value has not been formally evaluated and many physicians feel that not performing SIJ RFA in patients with negative SLBB may lead to withholding an effective treatment from patients. Thus, the standard practice is to proceed with SIJ RFA even with a negative SLBB because its prognostic value is not clear.

For the purpose of this study, all patients experiencing >50% pain relief after an intra articular SIJ injection of local anesthetic and corticosteroid but lasting less than 3 months and who wish to undergo SIJ RFA, as suggested by their treating physician, will be considered for inclusion in the study. Then, following general procedure, all patients will undergo a SLBB performed according to the previously described technique. The data from all the diaries will be collected to determine the rate of positive SLBBs among patients who had significant but not sustained pain relief from intraarticular SIJ injection. Then, all patients will proceed to SIJ RFA.

Recrutement:

Physicians will inform the research nurse when they meet a patient who had significant but non sustained pain relief after a SIJ injection and for which they consider SIJ RFA to be the next step in treatment.

The patient's file will be reviewed to confirm inclusion and exclusion criteria. All eligible patients will then be contacted by phone by a member of the research team to introduce them to the study protocol. A copy of the patient consent form will be sent by e-mail to patients who show interest in participating to the research project.

Patients will then be contacted again by phone the day prior to the procedure to answer any question and confirm their interest in participating to the study. Patients who wish to participate will be met by the research team on the day of their procedure and written consent will be obtained.

RF Procedure:

All procedures will be performed according to the standard of care for SIJ RFA at the Maisonneuve-Rosemont Hospital's Chronic Pain Clinic.

P-RF:

P-RF is performed using a conventional temperature-controlled RF generator (Diros Technology Inc's OWL, Markham, ON, Canada) generating monopolar and bipolar lesions at 85°C for 150 sec, with a 60 sec ramp time. Four, 18 Gauge 3-tined, 90 mm cannulas with an active tip of 10 mm (RF Trident; Diros Technology) will be used along with a four-output radiofrequency generator configured for quadripolar output.

Lesioning the sacral lateral branches:

* Under fluoroscopic guidance in the anteroposterior view, the C-arm is angulated cephalad in order to align the superior end plate of S1.
* Using a radiopaque marker, the superior border of the S1 posterior foramen is identified and the marker is placed slightly superior to this level, between the posterior foramen lateral border and the SIJ line. The overlying skin is marked with a sterile pen. The same marking procedure is accomplished, slightly inferior to the inferior border of the S3 posterior foramen. Using a sterile disposable ruler, a line connecting these two dots is drawn on the patient's skin and marked every 10 millimeters. The resulting line will typically be 55-60 mm long, and can be extended 5 mm in its superior and/or inferior part to allow sufficient space to place the uppermost and/or lowermost needle, allowing an inter-needle distance of 10 mm
* The skin is anesthetized with 1% lidocaine at each of the 10 mm marks, and four 3-tined RF needles are inserted under fluoroscopic guidance at the four uppermost marks. Intermittent fluoroscopy is used to ensure that the needles stay parallel to one another, perpendicular to the dorsal surface of the sacrum.
* Once contact with the dorsal surface of the sacrum is obtained, the C-arm is turned to obtain a lateral view to confirm that none of the needles went into the sacral foramen or landed on the posterior iliac crest (too shallow), and the tines are deployed.
* The four needles are connected to the four outputs of the quadripolaire radiofrequency generator. A motor stimulation test is carried out at each of the needles to ensure absence of motor stimulation in the lower limbs (2.0 V, 2 Hz), and 0,5 ml of 1% lidocaine is injected through the side port of each cannula. The RF energy is then delivered, making one quadripolar lesion. Then, the three uppermost cannulas are removed and two cannulas are inserted at the fifth and sixth mark, using the same technique as previously described, and two more sets of bipolar lesions are created, sequential (between needles 4 and 5, and then between 5 and 6) This procedure thus requires a total of 3 outputs of RF energy.

Lesioning the L5 dorsal ramus:

-Under fluoroscopic guidance in the anteroposterior view, the inflexion between the ala of the sacrum and the S1 superior articular process, is visualized. The RF needle is inserted from a point slightly lateral and inferior to the target until contact with the bone is made. Using a lateral view, the needle is confirmed to be no deeper than the anterior-posterior midline of the S1 superior articular process. The tines are deployed, and motor testing is performed to ensure absence of motor stimulation in the lower limb (2.0 V, 2 Hz). Sensory testing will not be performed as its benefits regarding clinical outcome are not endorsed by clinical guidelines. Then, 1 ml of 1% lidocaine is injected through the side port and the RF energy is delivered, creating a monopolar lesion.

Data collection

Baseline demographic data: Questionnaires will be answered by the patients in person, before the procedure.

Age, sex; Uni or bilateral lesioning; Average pain intensity over the last 7 days (Verbal Numeric scale score 0-10, where 0: no pain at all and 10: worse imaginable pain); Duration of pain (months); Smoking status; Opioid use and daily Oral Morphine Equivalent (OME); Fibromyalgia survey score (Widespread Pain Index + Symptom Severity Scale (Score /31)); Hospital Anxiety and Depression Score (HADS) Oswestry Disability Index score (ODI), Result (positive or negative) of the multi-site, multi-depth, sacral lateral branch block performed with 2% lidocaine. Positive= >50% pain relief for a duration of 2-24h, using a 36h pain diary evaluating pain intensity.

Follow up data

Patients will answer the questionnaires either in person at the Pain Clinic or from their home. In this case, patients will be contacted by phone at the time of the follow up to:

* Evaluate the average pain intensity over the last 7 days (VNS);
* Inform them that questionnaires were sent by e-mails and that they need to be completed and returned to the research team. Reminders will be sent after 2 and 4 weeks.

  1 month:
* Average pain intensity over the last 7 days (VNS 0-10). 3, 6 and 10 months:
* Average pain intensity over the last 7 days (VNS 0-10);
* Success (O/N), defined as >50% pain relief, compared to baseline;
* Patient Global Impression of Change Score (PGIC);
* ODI score;
* Opioid use over the last 7 days (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Low back pain caused by SIJ dysfunction lasting > 6 months:

  * Predominantly axial pain below the L5 vertebrae with an average daily Verbal Numercial Scale Score (VNS) >4;
  * >50% pain relief after a fluoroscopically guided intraarticular injection of local anesthetic and steroids in the SIJ but lasting less than 3 months. Injection performed in the last 6 months prior to enrollment.

Exclusion Criteria:

* Pregnancy

  * Spinal pathology that may impede recovery such as severe spondylolisthesis at L5/S1, severe scoliosis, or lumbar fusion;
  * Active radicular pain;
  * Worker's compensation;
  * Cognitive limitation or linguistic barrier making pain assessment through questionnaire impossible;
  * Implanted pacemaker or defibrillator;
  * Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for sacroiliac joint radio frequency ablation at the Maisonneuve-Rosemont Hospital's Chronic Pain Clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Success rate | 6 months
  proportion of patients reporting >50% pain relief

SECONDARY OUTCOMES:
Succes rate | 3 months
  proportion of patients reporting >50% pain relief
Succes rate | 1 month
  proportion of patients reporting >50% pain relief
Succes rate | 10 month
  proportion of patients reporting >50% pain relief
Change in Pain score | 1 month
  mean change in pain score using a verbal numeric pain scale of 0-10 (0: no pain, 10: worse imaginable pain)
Change in Pain score | 3 month
  mean change in pain score using a verbal numeric pain scale of 0-10 (0: no pain, 10: worse imaginable pain)
Change in Pain score | 6 month
  mean change in pain score using a verbal numeric pain scale of 0-10 (0: no pain, 10: worse imaginable pain)
Chang in Pain score | 10 month
  mean change in pain score using a verbal numeric pain scale of 0-10 (0: no pain, 10: worse imaginable pain)
Impact on disability | 3 months
  change in the Owestry Disability Index (scale 0-100 where 0: minimal disability, 100: crippled)
Impact on disability | 6 months
  change in the Owestry Disability Index (scale 0-100 where 0: minimal disability, 100: crippled)
Impact on disability | 10 months
  change in the Owestry Disability Index (scale 0-100 where 0: minimal disability, 100: crippled)
Impact on improvement | 3 months
  Patient global impression of change scale score (scale of 1-7 where 1: very much improved, 7: very much worse
Impact on improvement | 6 months
  Patient global impression of change scale score (scale of 1-7 where 1: very much improved, 7: very much worse
Impact on improvement | 10 months
  Patient global impression of change scale score (scale of 1-7 where 1: very much improved, 7: very much worse
Opioid use | 3 months
  determine the impact of the intervention on the opioid daily dose(determined by calculating Oral Morphine Equivalent)(mg)
Opioid use | 6 months
  determine the impact of the intervention on the opioid daily dose (determined by calculating Oral Morphine Equivalent)(mg)
Opioid use | 10 months
  determine the impact of the intervention on daily opioid dose (determined by calculating Oral Morphine Equivalent)(mg)

OTHER OUTCOMES:
analgesia from sacral lateral branch block | baseline
  determine the proportion of patients reporting >50% pain relief after a sacral lateral branch block, among patients with presumed pain from sacroiliac joint
Success rate | 3 months
  proportion of patients reporting >50% pain relief in patients who had a negative sacral lateral branch block, compared to patients with a positive sacral lateral branch block
Success rate | 6 months
  proportion of patients reporting >50% pain relief in patients who had a negative sacral lateral branch block, compared to patients with a positive sacral lateral branch block
Success rate | 10 months
  proportion of patients reporting >50% pain relief in patients who had a negative sacral lateral branch block, compared to patients with a positive sacral lateral branch block

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada